CLINICAL TRIAL: NCT03443557
Title: Effects of Oral Nutrition Supplement in Thai Malnourished Patients : A Cross-sectional Nutrition Day Survey
Brief Title: Effects of Oral Nutrition Supplement in Thai Malnourished Patients
Status: Completed | Type: Observational
Sponsor: Pierre Singer (Other)
Responsible Party: Sponsor-Investigator, Pierre Singer, Professor, Rabin Medical Center
Organization: Rabin Medical Center (Other)
Other Study IDs: 0829-17-RMC
Record Dates: First submitted 2018-02-18; First posted 2018-02-23 (Actual); Last update posted 2018-03-13 (Actual); Status verified 2018-03

CONDITIONS: Malnourished; Hospitalized
Keywords: Oral nutrition supplement; malnutrition; mortality
MeSH Terms: conditions — Malnutrition

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Cross-Sectional
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- oral nutrition supplement group: hospitalized malnourished patients who were received oral nutrition supplement during hospital course
  Interventions: Other: oral nutrition supplement
- control group: hospitalized malnourished patients who were received only hospital food during hospital course

INTERVENTIONS:
Other: oral nutrition supplement — receiving prescription of oral nutrition supplement during hospitalization
  Groups: oral nutrition supplement group

SUMMARY:
A retrospective study based on Thai data from Nutrition Day study (nD). Comparing clinical outcome between malnourished patients who were prescribed oral nutrition supplement along with hospital diet and those without oral nutrition supplement.

DETAILED DESCRIPTION:
Prevalence of malnutrition in hospitalized patients varies from 30-70% depend on category of patients recruited. Adverse effects of malnutrition include increase of infection complication, increase hospital length of stay, and increase mortality. Prescription of oral nutrition supplement (ONS) have been proved to provide patients more calorie and protein intake and can improve patients' outcome.

Despite the proved benefits of oral nutrition supplement(ONS), prescription of it in Thai hospitalized patients are far less than it should. The main reason of this under-practice is the limitation of health policies which considered ONS as an optional from main meals. Additional cost for ONS has to be paid by patients themselves, therefore the patients who have no willing to pay usually refuse to receive ONS. Unawareness of physician regarding its benefits is also a problem. In order to convince Thai authorities to allow for reimbursement of ONS and encourage prescription of ONS among physicians, an evidence based benefits of ONS in large Thai population is needed.

The nD study was a single-day, population-based, standardized, multinational, cross-sectional audit and was performed worldwide, includes Thailand, in hospitals, nursing homes and intensive care units performing since 2006 to present. Every year, registered hospitals survey their patients regarding nutritional status, nutritional support. A follow-up for clinical outcome are perform at 30 days after the first survey, include mortality, readmission. This study will based on data of Thai patients collected from nD study during 2006-2016.

ELIGIBILITY:
Inclusion Criteria:

* Age 18 years old and above
* identified as malnourished or at risk

Exclusion Criteria:

* terminally ill patients
* receiving concomitant enteral tube feeding and/or supplemental parenteral nutrition

Min Age: 18 Years | Sex: All
Age Groups: Adult, Older Adult
Study Population: Thai hospitalized patients
Sampling Method: Non-Probability Sample
Enrollment: 500 (Actual)
Dates: Start 2006-01-01 (Actual); Primary Completion 2016-11-30 (Actual); Study Completion 2016-12-31 (Actual)

PRIMARY OUTCOMES:
30-day mortality | 30 days
  dead rate at 30 days after study date will be extracted from hospital medical record by hospital staff

SECONDARY OUTCOMES:
Discharge rate | 30 days
  Discharge status at 30 day will be extracted from hospital medical record by hospital staff
Hospital length of stay | 30 days
  Hospital length of stay will be extracted from hospital medical record by hospital staff
Re-admission rate | 30 days
  Re-admission rate will be extracted from hospital medical record by hospital staff

OTHER OUTCOMES:
prevalence of oral nutrition supplement prescription in Thai hospitalized patients | 10 years
  prevalence of oral nutrition supplement prescription in Thai hospitalized patients

CONTACTS AND LOCATIONS:
Overall Officials: Pierre Singer, Professor, Principal Investigator — Rabin Medical Center
Locations (1):
- Rabin medical center, Petah Tikva, Israel

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- [Background] Milne AC, Potter J, Vivanti A, Avenell A. Protein and energy supplementation in elderly people at risk from malnutrition. Cochrane Database Syst Rev. 2009 Apr 15;2009(2):CD003288. doi: 10.1002/14651858.CD003288.pub3. PMID 19370584
- [Background] Philipson TJ, Snider JT, Lakdawalla DN, Stryckman B, Goldman DP. Impact of oral nutritional supplementation on hospital outcomes. Am J Manag Care. 2013 Feb;19(2):121-8. PMID 23448109
- [Background] Norman K, Kirchner H, Freudenreich M, Ockenga J, Lochs H, Pirlich M. Three month intervention with protein and energy rich supplements improve muscle function and quality of life in malnourished patients with non-neoplastic gastrointestinal disease--a randomized controlled trial. Clin Nutr. 2008 Feb;27(1):48-56. doi: 10.1016/j.clnu.2007.08.011. Epub 2007 Oct 25. PMID 17964008